CLINICAL TRIAL: NCT04770207
Title: Intra-tumor Injection of Drug-eluting Microspheres Loading With Chemodrug Plus Checkpoint Inhibitors and/or IL2 for Treatment of Advanced Solid Tumors
Brief Title: Intra-tumor Injection of Drug-eluting Microspheres With Multiple Drugs
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZITDEB-010
Record Dates: First submitted 2020-12-02; First posted 2021-02-25 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma; Solid Tumor, Adult
Keywords: Hepatocellular Carcinoma; Lung Cancer; Solid Tumors; Drug-eluting Beads; IL2; Kytruda; Opdivo; Imfinza; Atezolizumab; Ipilimumab;; Treprizolizumab; Tirelizumab; Carellizumab; Sintilimab;; Sugemalimab；Adebrelimab；Envafolimab；Cadonilimab；; Bevacizumab; Ramucirumab
MeSH Terms: conditions — Carcinoma, Hepatocellular; Lung Neoplasms | interventions — cyclopropapyrroloindole; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Drug-eluting beads loaded with various drugs including IL2, kytruda, imfinzi, yevoy, bevacizumag, or/and ramucirumab, doxorubicin/idarubicin are injected into solid tumors under CT guidance according to appropriate treatment strategy, once per 3-6 weeks, and the safety and efficacy will be evaluated by guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: DC-Beads loading with Chemodrug/IL2/PD1/CTLA4 antibodies (Experimental): Intra-tumor injection of above drugs for patients with previous treatment with PDL1 antibody and relapsed.
  Interventions: Drug: Injection of drug-eluting microspheres with multiple drugs into solid tumors
- Group 2: DC-Beads loading with Chemodrug/IL2/PDL1/CTLA4 antibodies (Experimental): Intra-tumor injection of above drugs for patients with previous treatment with PD1 antibody and relapsed.
  Interventions: Drug: Injection of drug-eluting microspheres with multiple drugs into solid tumors
- Group 3: DC-Beads loading with Chemodrug/IL2/PD1/PDL1/CTLA4 antibodies (Experimental): Intra-tumor injection of above drugs for patients with previous heavily treated with PD1/PDL1/CTLA4 antibodies and relapsed.
  Interventions: Drug: Injection of drug-eluting microspheres with multiple drugs into solid tumors

INTERVENTIONS:
Drug: Injection of drug-eluting microspheres with multiple drugs into solid tumors — Under the guidance of CT, puncture fine needle was used to inject drug-eluting microspheres loading with multiple drugs into the tumor
  Other Names: Checkpoint inhibitor (CPI) such as Keytruda plus chemodrug

SUMMARY:
To study the safety and clinical effect of injection of drug-eluting microspheres with multiple chemodrug and/or protein drugs into advanced solid tumors.

DETAILED DESCRIPTION:
Drug-eluting microspheres such as DC-beads will be loaded with IL2, PD1/PDL1/CTLA4 antibody, or /and VEGF/VEGFR antibody with or without doxorubicin/idarubicin for various time and injected into tumors under CT guidance. Side effects and treatment efficacy after injection of drug-eluting microspheres into malignant tumors will be assessed according to RICEST1.1 standard.

ELIGIBILITY:
Inclusion Criteria:

* Solid advanced malignant tumors
* Age between18 and 99 years
* Life expectancy is greater than three months

Exclusion Criteria:

* Benign tumor
* Life expectancy is less than three months
* Serious medical comorbidity
* Others

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2035-11-01 (Estimated)

PRIMARY OUTCOMES:
Assessing safety and treatment efficacy on intra-tumor injection of DEB for advanced tumors | up to 36 months
  Assessing incidence of side effects and primary clinical response of the intra-tumor injection of DEB in advanced solid cancers, including CR, PR, SD, and PD.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borde T, Laage Gaupp F, Geschwind JF, Savic LJ, Miszczuk M, Rexha I, Adam L, Walsh JJ, Huber S, Duncan JS, Peters DC, Sinusas A, Schlachter T, Gebauer B, Hyder F, Coman D, van Breugel JMM, Chapiro J. Idarubicin-Loaded ONCOZENE Drug-Eluting Bead Chemoembolization in a Rabbit Liver Tumor Model: Investigating Safety, Therapeutic Efficacy, and Effects on Tumor Microenvironment. J Vasc Interv Radiol. 2020 Oct;31(10):1706-1716.e1. doi: 10.1016/j.jvir.2020.04.010. Epub 2020 Jul 17. PMID 32684417
- [Background] Binder S, Lewis AL, Lohr JM, Keese M. Extravascular use of drug-eluting beads: a promising approach in compartment-based tumor therapy. World J Gastroenterol. 2013 Nov 21;19(43):7586-93. doi: 10.3748/wjg.v19.i43.7586. PMID 24282349
- [Background] Baur J, Ritter CO, Germer CT, Klein I, Kickuth R, Steger U. Transarterial chemoembolization with drug-eluting beads versus conventional transarterial chemoembolization in locally advanced hepatocellular carcinoma. Hepat Med. 2016 Jun 20;8:69-74. doi: 10.2147/HMER.S105395. eCollection 2016. PMID 27382341
- [Background] Malagari K. Drug-eluting particles in the treatment of HCC: chemoembolization with doxorubicin-loaded DC Bead. Expert Rev Anticancer Ther. 2008 Oct;8(10):1643-50. doi: 10.1586/14737140.8.10.1643. PMID 18925855
- [Background] Rossi SM, Murray T, McDonough L, Kelly H. Loco-regional drug delivery in oncology: current clinical applications and future translational opportunities. Expert Opin Drug Deliv. 2021 May;18(5):607-623. doi: 10.1080/17425247.2021.1856074. Epub 2020 Dec 16. PMID 33253052
- [Background] Fuchs K, Duran R, Denys A, Bize PE, Borchard G, Jordan O. Drug-eluting embolic microspheres for local drug delivery - State of the art. J Control Release. 2017 Sep 28;262:127-138. doi: 10.1016/j.jconrel.2017.07.016. Epub 2017 Jul 11. PMID 28710006